CLINICAL TRIAL: NCT00250029
Title: Gene Expression Analysis of Patients With Metastatic Colorectal Cancer Receiving Oxaliplatin Based Chemotherapy
Brief Title: Gene Expression Analysis of Patients With Metastatic Colorectal Cancer Receiving Oxaliplatin Based Chemotherapy Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0104C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2010-04

CONDITIONS: Colonic Diseases; Cancer
Keywords: Colorectal Cancer; Pilot Study; Oxaliplatin
MeSH Terms: conditions — Colonic Diseases; Neoplasms; Colorectal Neoplasms | interventions — Oxaliplatin; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered at the dose of 130 mg/m2 given as a 2 hour intravenous infusion on day 1 of a three week cycle, prior to the 1st dose of capecitabine. 5-HT3 antagonists with or without dexamethasone premedication are strongly recommended. Oxaliplatin may be infused either through a peripheral vein or a central venous line. The infusion lines must be adequately flushed with 5% dextrose solution (D5W) between oxaliplatin infusion & the administration of any other drug.
  Capecitabine is to be administered orally within 30 mins. after the end of a meal. Tablets should be swallowed with approximately 200 mL water (not fruit juices). The first dose of each cycle will be administered as the evening dose on day 1 & the last dose of each cycle is scheduled the morning of day 15, followed by a 7 day rest period. This provides for a total of 28 single doses per cycle over 15 calendar days.
  Other Names: XELOX (oxaplatin+capecitabine)

SUMMARY:
1.1 To collect pathological tumor specimens of patients with metastatic colorectal cancer in a prospective fashion for correlative studies of response to an oxaliplatin based chemotherapy regimen.

1.2 To determine a gene expression profile that predicts response to an oxaliplatin based chemotherapy regimen in this cohort of patients.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized trial of oxaliplatin and capecitabine. Patients that are placed on other studies that utilize the same chemotherapy regimen can enter this study. Those patients will be treated according to the clinical study on which they have been entered. For patients not on another clinical trial, the treatment outlined below should be followed.

ELIGIBILITY:
Inclusion Criteria:

* All patients, >18 years of age, with metastatic/recurrent colorectal cancer are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count > 100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* The patient must agree to a biopsy of a sample of tumor for correlative studies.
* The patient is an appropriate candidate for oxaliplatin/capecitabine based chemotherapy.
* The patient must have measurable disease.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Patients may not have received oxaliplatin previously.
* Patients with a prior unanticipated severe reaction to fluoropyrimidine therapy, or known dihydropyrimidine dehydrogenase (DPD) deficiency, or known hypersensitivity to platinum compounds or any of the components of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04; Primary Completion 2005-09 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To collect pathological tumor specimens of patients with metastatic colorectal cancer in a prospective fashion for correlative studies of response to an oxaliplatin based chemotherapy regimen | The cycle length is 3 weeks, consisting of 2 weeks of capecitabine treatment followed by 1 week without treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (4):
- United States (4):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Lovelace Sandia Health Systems Dept of Hematology, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Veterans Administration Health Care System, Albuquerque, New Mexico